CLINICAL TRIAL: NCT01015742
Title: Evaluation of Benefit and Side Effects of Double Umbilical Cord Blood Units Stem Cell Transplantation in Hematologic Malignancies
Brief Title: Unrelated Double Umbilical Cord Blood Units Transplantation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HORCSCT-0902
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoblastic, Acute; Leukemia, Myeloid, Chronic
Keywords: AML; ALL; CML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Stem cell Transplant using two unrelated umbilical cord blood units.
  Interventions: Drug: Stem cell Transplantation

INTERVENTIONS:
Drug: Stem cell Transplantation — Busulfan: 3.2 mg/kg IV daily on days -7 to -4
  Cyclophosphamide : 60 mg/m² daily on days -3 to -2
  Rabbit Thymoglobulin 2.5mg/kg IV daily on days -3 to -2
  Cyclosporin will begin on day -2 (IV or oral) for at least 180 days. Target trough level for cyclosporin is 200 ng/ml. In the absence of GVHD, Cyclosporin tapering will begin on day +90
  Methyl prednisolone (1mg/kg/d IV) will begin on day -2 to +7 and then 0.5mg/kg until +14 posttransplant.

SUMMARY:
The purpose of this study is to determine the safety and feasibility of unrelated double umbilical cord blood units Transplantation in patients with haematological malignancies using Antithymocyte Globulin Cyclophosphamide, busulfan as conditioning and cyclosporin, methylprednisolone as GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Hematologically & Histologically confirmed acute lymphoblastic or acute and chronic myeloid leukemia in Remission
* Aged 1 year to 50 years
* Absence of HLA compatible related or other related donor.
* Availability of suitable UCB units.
* karnofsky performance score (> 12 yr) or lansky play performance(<12 yr) : 80- 100
* Adequate renal function defined as:Serum creatinine <1.5 x normal,
* Adequate liver function defined as:Total bilirubin <1.5 x normal, or SGOT (AST) or SGPT (ALT) <3.0 x normal
* Adequate cardiac function defined as: Ejection fraction >50% by echocardiogram.
* Adequate pulmonary function defined as:Uncorrected DLCO 50% by pulmonary function test.For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air

Exclusion Criteria:

* Age: < 1year or > 50 year
* Patients with an available 5-6/6 HLA-A, -B, -DRB1 matched sibling or other related donor
* karnofsky performance score (> 12 yr) or lansky play performance(<12 yr) < 80
* HIV positive patients.
* Female patients who are pregnant or breast feeding
* Life expectancy severely limited by diseases of vital organs other than the disease indication for transplant
* Serious concurrent untreated infection e.g. active tuberculosis, mycoses or viral infection
* Serious psychiatric/ psychological disorders
* Absence of /inability to provide informed consent
* Clinical or Paraclinical evidence of CNS or PNS involvement

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
To determine the Benefit and Side Effects of Double Umbilical Cord Blood Units Stem Cell Transplantation in Hematologic Malignancies | Until end of study

SECONDARY OUTCOMES:
Neutrophil and platelet engraftment | 1 year
Severity of acute graft-vs-host disease(GvHD | 1 year
Early transplant related mortality | 100 days
Overall and disease free survival at one years | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amir Ali Hamidieh, MD, Principal Investigator — Hematology-Oncology and SCT Research Center
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Tehran Province, Iran